CLINICAL TRIAL: NCT01475786
Title: A Phase II, Double-Blind, Randomized, Placebo-Controlled, Multicenter Study to Assess the Safety and Efficacy of Engensis (VM202) in Subjects With Painful Diabetic Peripheral Neuropathy
Brief Title: Safety and Efficacy Study for the Treatment of Painful Diabetic Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Helixmith Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VMDN-002
Record Dates: First submitted 2011-11-15; First posted 2011-11-21 (Estimated); Results first posted 2023-07-03 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-08

CONDITIONS: Painful Diabetic Neuropathies
Keywords: nerve pain; diabetic nerve pain; throbbing; burning; painful feet; tingling; numbness; Engensis (VM202)
MeSH Terms: conditions — Diabetic Neuropathies; Neuralgia; Paresthesia; Hypesthesia | interventions — Genetic Therapy; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low Dose 16mg Engensis (VM202) and Placebo (Active Comparator): intramuscular injections in each calf for a total of 16mg Engensis (VM202): Day 0 - 32 injections / calf 16 injections of 0.5mL of VM202 / calf - (4 mg of VM202 / calf) and 16 injections of normal saline 0.5mL / calf Day 14 - 32 injections / calf and 16 injections of normal saline 0.5mL / calf 16 injections of 0.5mL of VM202 / calf - (4 mg of VM202 / calf)
  Interventions: Biological: Low Dose: 16 mg Engensis (VM202); Other: Control- Placebo (normal saline)
- High Dose 32mg Engensis (VM202) (Active Comparator): Day 0 - 32 injections of 0.5mL of VM202 / calf (8 mg of VM202 / calf) Day 14 - 32 injections of 0.5mL of VM202 / calf (8 mg of VM202 / calf) For a total of 32mg VM202
  Interventions: Biological: High Dose: 32 mg Engensis (VM202)
- Control - Placebo (normal saline) (Placebo Comparator): 32 injections / calf of 0.5 mL normal saline at Day 0 and Day 14
  Interventions: Other: Control- Placebo (normal saline)

INTERVENTIONS:
Biological: Low Dose: 16 mg Engensis (VM202) — Subjects in the Low Dose Group (8mg VM202 / leg) will receive the following intramuscular injections in each calf:
  Day 0 - 32 injections / calf:
  • 16 injections of 0.5mL of VM202 / calf - (4 mg of VM202 / calf)
  Day 14 - 32 injections / calf:
  • 16 injections of 0.5mL of VM202 / calf - (4 mg of VM202 / calf)
  Other Names: Gene Therapy
  Arms: Low Dose 16mg Engensis (VM202) and Placebo
Biological: High Dose: 32 mg Engensis (VM202) — Subjects in the High Dose Group (16 mg VM202 / leg) will receive the following intramuscular injections in each calf:
  Day 0
  • 32 injections of 0.5mL of VM202 / calf (8 mg of VM202 / calf)
  Day 14
  • 32 injections of 0.5mL of VM202 / calf (8 mg of VM202 / calf)
  Other Names: Gene Therapy
  Arms: High Dose 32mg Engensis (VM202)
Other: Control- Placebo (normal saline) — subjects will receive thirty-two (32) 0.5 mL injections of normal saline on Day 0 and Day 14.
  Other Names: Normal saline
  Arms: Control - Placebo (normal saline); Low Dose 16mg Engensis (VM202) and Placebo

SUMMARY:
The purpose of this study is to determine if Engensis (VM202) is safe and effective in treating painful diabetic neuropathy.

DETAILED DESCRIPTION:
Peripheral neuropathy is a serious complication of diabetes. This form of neuropathy carries a high risk of pain, trophic changes and autonomic dysfunction. There is currently no effective treatment for diabetic neuropathy, and good glycemic control is the only way to minimize the risk of occurrence. Clearly, it would be desirable to prevent, impede, or reverse the disrupting and often life-threatening manifestations of peripheral neuropathy by stimulating growth or regeneration of peripheral nerve axons.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years to ≤ 75 years
* Documented history of Type I or II diabetes with current treatment control (glycosylated hemoglobin A1c of ≤ 10.0% at Screening) and currently on oral medication and/or insulin
* Diagnosis of painful diabetic peripheral neuropathy in both lower extremities
* Lower extremity pain for at least 6 months
* Visual analog scale (VAS) score of ≥ 40 mm at Initial Screening (0 mm = no pain - 100 mm very severe pain)
* Symptoms from the Brief Pain Neuropathy Screening (BPNS) is ≤ 5 point difference between legs at Initial Screening
* The average daily pain intensity score of the Daily Pain and Sleep Interference Diary completed after medication wash-out is ≥ 4 with a standard deviation ≤ 2
* The physical examination component of the Michigan Neuropathy Screening Instrument Score (MNSI) is ≥ 3 at Screening
* Stable treatment of diabetes for at least 3 months with no anticipated changes in medication regimen, and no new symptoms associated with diabetes
* If female of childbearing potential, negative urine pregnancy test at screening and using acceptable method of birth control during the study

Exclusion Criteria:

* Peripheral neuropathy caused by condition other than diabetes
* Other pain more severe than neuropathic pain
* Progressive or degenerative neurological disorder
* Myopathy
* Inflammatory disorder of the blood vessels (inflammatory angiopathy, such as Buerger's disease)
* Active infection
* Chronic inflammatory disease (e.g., Crohn's disease, rheumatoid arthritis)
* Positive HIV or HTLV at Screening
* Active Hepatitis B or C as determined by Hepatitis B core antibody (HBcAB), antibody to Hepatitis B antigen (IgG and IgM; HbsAb), Hepatitis B surface antigen (HBsAg) and Hepatitis C antibodies (Anti-HCV) at Screening
* Subjects with known immunosuppression or currently receiving immunosuppressive drugs, chemotherapy or radiation therapy
* Stroke or myocardial infarction within last 3 months
* Ophthalmologic conditions pertinent to proliferative retinopathy or conditions that preclude standard ophthalmologic examination
* Specific laboratory values at Screening including: Hemoglobin < 8.0 g/dL, WBC < 3,000 cells per microliter, platelet count <75,000/mm3, Creatinine > 2.0 mg/dL; AST and/or ALT > 3 times the upper limit of normal or any other clinically significant lab abnormality which in the opinion of the investigator should be exclusionary
* Uncontrolled hypertension as defined as sustained systolic blood pressure (SBP) > 200 mmHg or diastolic BP (DBP) > 110 mmHg at Screening
* Patients with a recent history (< 5 years) of or new screening finding of malignant neoplasm except basal cell carcinoma or squamous cell carcinoma of the skin (if excised and no evidence of recurrence); patients with family history of colon cancer in any first degree relative are excluded unless they have undergone a colonoscopy in the last 12 months with negative findings
* Subjects requiring > 81 mg daily of acetylsalicylic acid; If ≥ 81 mg are taken at screening, subjects may be enrolled if willing/able to switch to another medication
* Use of any opioids; subjects may be enrolled if willing and able to discontinue use of these drugs 14 days prior to starting the 7 Day Daily Pain and Sleep Interference Diary and refrain from taking these drugs for the duration of the study
* Subjects requiring regular COX-2 inhibitor drug(s) or non-specific COX-1/COX-2 inhibiting drugs, or high dose steroids (excepting inhaled steroids).Subjects may be enrolled if willing/able to undergo medication wash-out prior to the first dosing and to refrain from taking these drugs for the duration of the study;
* Major psychiatric disorder in within last 6 months
* Body mass index (BMI) > 45 kg/m2 at Screening
* Any lower extremity amputation
* Use of an investigational drug or treatment in past 6 months
* Unable or unwilling to give informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2012-08; Primary Completion 2014-03-12 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jack Kessler, MD, Principal Investigator — Northwestern University
Locations (17):
- United States (13):
  - Diablo Clinical Research, Walnut Creek, California
  - Compass Research, Orlando, Florida
  - Palm Beach Neurological Center, Palm Beach Gardens, Florida
  - Northwestern University, Chicago, Illinois
  - Beth Israel Deaconess, Boston, Massachusetts
  - The Neurosciences Institute Albany Medical College, Albany, New York
  - Mount Sinai Medical Center, New York, New York
  - University of Oklahoma Harold Hamm Diabetes Center, Oklahoma City, Oklahoma
  - Houston Neurocare, Houston, Texas
  - The Methodist Hospital, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - East Virginia Medical School Strelitz Diabetes Center, Norfolk, Virginia
  - Rainier Clinical Research, Seattle, Washington
- South Korea (4):
  - Seoul National University Bundang Hospital, Seongnam, Bundang-gu
  - Yonsei University College of Medicine Severance Hospital, Seoul, Seodaemun-gu
  - Sejong General Hospital, Bucheon-si, Sosa-gu
  - The Catholic University of Korea Youido St. Mary's Hospital, Seoul, Yeongdeungpo-gu

REFERENCES:
- [Result] Kessler JA, Smith AG, Cha BS, Choi SH, Wymer J, Shaibani A, Ajroud-Driss S, Vinik A; VM202 DPN-II Study Group. Double-blind, placebo-controlled study of HGF gene therapy in diabetic neuropathy. Ann Clin Transl Neurol. 2015 May;2(5):465-78. doi: 10.1002/acn3.186. Epub 2015 Mar 5. PMID 26000320

RESULTS

PARTICIPANT FLOW:
Groups:
- High Dose 32mg Engensis (VM202): Subjects in the High Dose Group (16 mg VM202 / leg) received the following intramuscular injections in each calf for a total of 32 mg Engensis (VM202):
  Day 0 - 32 injections of 0.5 mL of VM202 / calf (8 mg of VM202 / calf)
  Day 14 - 32 injections of 0.5 mL of VM202 / calf (8 mg of VM202 / calf) For a total of 32mg VM202
- Low Dose 16mg Engensis (VM202) and Placebo: Subjects in the Low Dose Group (8 mg/leg) received the following intramuscular injections in each calf for a total of 16mg Engensis (VM202):
  : Day 0 - 32 injections / calf 16 injections of 0.5mL of VM202 / calf - (4 mg of VM202 / calf) and 16 injections of Placebo 0.5mL / calf
  Day 14 - 32 injections / calf 16 injections of 0.5mL of VM202 / calf - (4 mg of VM202 / calf) and 16 injections of Placebo 0.5mL / calf
- Control - Placebo (Normal Saline): Subjects in the Placebo Group received 32 injections / calf of 0.5 mL Placebo on Day 0 and Day 14
Period: Overall Study
Arm/Group | High Dose 32mg Engensis (VM202) | Low Dose 16mg Engensis (VM202) and Placebo | Control - Placebo (Normal Saline)
Started | 43 | 40 | 21
Completed | 41 | 36 | 19
Not Completed | 2 | 4 | 2
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Subject discontinued prior to study treatment | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Subjects in the intent to treat (ITT) population were those who were randomized and received study treatments
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose 32mg Engensis (VM202) | Low Dose 16mg Engensis (VM202) and Placebo | Control - Placebo (Normal Saline) | Total
Number analyzed (Participants) | 42 | 40 | 21 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (10.2) | 60.2 (7.2) | 60.5 (8.3) | 60.4 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 6 | 26
  Male | 33 | 29 | 15 | 77
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 6 | 5 | 6 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 7 | 2 | 12
  White | 32 | 27 | 12 | 71
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 42 | 40 | 21 | 103

OUTCOME MEASURES:

1. Primary Outcome: The Primary Study Endpoint Was the Change in Average 24-hour Pain Score From Baseline to the 6-month Follow-up.
Description: The difference in the mean change of the 24 hour pain score was compared between the treatment groups and the placebo arm to determine treatment effect. The average pain scores were obtained from the Daily Pain and Sleep Interference Diary (recorded daily by subjects for 7 days during Screening prior to the first round of injections and again, before the 6 month follow-up). Subjects rated their 24-hor daily pain intensity according to the 11-point numerical rating scale from 0 (no pain) to 10 (worst possible pain).
Time Frame: seven (7) days before 9 Month visit
Population: The Efficacy population included all subjects who received the correct dose of study drug based on the randomization schedule at both Days 0 and 14, have the Day 180 assessment, and did not have any protocol violations or major deviations
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- High Dose 32mg Engensis (VM202): Subjects in the High Dose Group (16 mg VM202 / leg) received the following intramuscular injections in each calf for a total of 32 mg Engensis (VM202):
  Day 0: 32 injections of 0.5 mL of VM202 / calf (8 mg of VM202 / calf)
  Day 14: 32 injections of 0.5 mL of VM202 / calf (8 mg of VM202 / calf) For a total of 32mg VM202
- Low Dose 16mg Engensis (VM202) and Placebo: Subjects in the Low Dose Group (8 mg/leg) received the following intramuscular injections in each calf for a total of 16mg Engensis (VM202):
  : Day 0: 32 injections / calf 16 injections of 0.5mL of VM202 / calf - (4 mg of VM202 / calf) and 16 injections of Placebo 0.5mL / calf
  Day 14: 32 injections / calf 16 injections of 0.5mL of VM202 / calf - (4 mg of VM202 / calf) and 16 injections of Placebo 0.5mL / calf
Arm/Group | High Dose 32mg Engensis (VM202) | Low Dose 16mg Engensis (VM202) and Placebo | Control - Placebo (Normal Saline)
Number analyzed (Participants) | 36 | 31 | 17
units on a scale | -1.94 (1.96) | -2.78 (2.23) | -1.59 (1.89)

ADVERSE EVENTS:
Time Frame: Baseline (Day 0) to Day 270
Arm/Group | High Dose 32mg Engensis (VM202) | Low Dose 16mg Engensis (VM202) and Placebo | Control - Placebo (Normal Saline)
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/39 | 0/21
Serious Adverse Events (participants affected / at risk) | 4/43 | 3/39 | 3/21
Other Adverse Events (participants affected / at risk) | 33/43 | 22/39 | 13/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High Dose 32mg Engensis (VM202) (N=43) | Low Dose 16mg Engensis (VM202) and Placebo (N=39) | Control - Placebo (Normal Saline) (N=21)
Left ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0
Omental infarction (Gastrointestinal disorders) | 0 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Asthma (Immune system disorders) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Localised infection (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Spontaneous cerebrospinal fluid leak (Nervous system disorders) | 1 | 0 | 0
Drug abuse (Psychiatric disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | High Dose 32mg Engensis (VM202) (N=43) | Low Dose 16mg Engensis (VM202) and Placebo (N=39) | Control - Placebo (Normal Saline) (N=21)
Localised infection (Infections and infestations) | 4 | 3 | 1
Sinusitis (Infections and infestations) | 0 | 5 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 2
Bronchitis (Infections and infestations) | 0 | 1 | 2
Nasopharyngitis (Infections and infestations) | 3 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 1 | 1
Ligament sprain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 3
Nausea (Gastrointestinal disorders) | 3 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 3 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 2 | 0
Cataract (Eye disorders) | 2 | 1 | 0
Chest pain (General disorders) | 2 | 1 | 0
Oedema peripheral (General disorders) | 2 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Hypertension (Vascular disorders) | 2 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2012-08-01): https://cdn.clinicaltrials.gov/large-docs/86/NCT01475786/Prot_000.pdf
  • Statistical Analysis Plan (2014-04-09): https://cdn.clinicaltrials.gov/large-docs/86/NCT01475786/SAP_001.pdf